CLINICAL TRIAL: NCT03188874
Title: Clinical AML Registry and Biomaterial Database of the Study Alliance Leukemia (SAL)
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: SAL-AML-REG-BIO
Record Dates: First submitted 2017-03-01; First posted 2017-06-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — bone marrow and peripher blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a registry study in adult patients with newly diagnosed or refractory/relapsed acute myeloid leukemia.

Investigator's sites: 51 sites in Germany.

Primary objectives:

* Identification of epidemiological data on AML: age, prognostic factors and subgroup distributions. Incidence and age distribution are compared with the data of population-related tumor registry.
* Evaluation of the most important patient-relevant clinical endpoints (outcomes): relapse-free survival (RFS) / time to relapse (TTR), calculation of cumulative incidence of relapse (CIR) and overall survival (OS)
* Documentation of treatment strategy

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* AML according to the WHO (World Health Organization) diagnostic criteria, including acute promyelocytic leukemia
* Age ≥ 18 years. There is no upper age limit.
* Signed written informed consent

Exclusion Criteria:

* there are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly-diagnosed AML, including acute promyelocytic leukemia (APL)
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2010-09; Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiological parameters | 10 years
  Epidemiological parameters
Relapse free survival (RFS) | 10 years
  Relapse free survival
Time to relapse (TTR), | 10 years
  Time to relapse (TTR),
Overall Survival (OS) | 10 years
  Overall Survival (OS)
cumulative incidence of relapse (CIR) | 10 years
  cumulative incidence of relapse (CIR)

SECONDARY OUTCOMES:
Complete Remission (CR) | yearly follow up 10 years
  Complete Remission
Treatment related mortality (TRM) | yearly follow up 10 years
  Treatment related mortality
Therapy-associated morbidity | yearly follow up 10 years
  grade IV toxicities
Recording and evaluating the quality of therapy and diagnosis | 10 years
  Recording and evaluating the quality of therapy and diagnosis
Validation of published prognostic factors at the registry cohort and the search for new possible prognostic factors | 10 years
  Validation of published prognostic factors at the registry cohort and the search for new possible prognostic factors
Recording and describing new forms of therapy and new supportive measures | 10 years
  Recording and describing new forms of therapy and new supportive measures

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof. Dr., Study Director — Universitätsklinikum Carl Gustav Carus
Locations (51):
- Germany (51):
  - Klinikum Mittelbaden, Baden-Baden, Baden-Wurttemberg
  - Universtitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Diakonie-Klinikum, Schwäbisch Hall, Baden-Wurttemberg
  - Kliniken Sindelfingen-Böblingen gGmbH, Sindelfingen, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart, Baden-Wurttemberg
  - Rems-Murr-Klinikum Winnenden, Winnenden, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Sozialstiftung Bamberg, Bamberg, Bavaria
  - Klinikum Bayreuth GmbH, Bayreuth, Bavaria
  - MVZ Klinikum Coburg GmbH, Coburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus, Brandenburg
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder), Brandenburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Klinikum Fulda / MVZ Osthessen GmbH, Fulda, Hesse
  - Universitätsklinikum Gießen und Marburg, Marburg, Hesse
  - Dr. Horst Schmidt Kliniken GmbH, Wiesbaden, Hesse
  - St. Bernward Krankenhaus Hildesheim, Hildesheim, Lower Saxony
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme), Lower Saxony
  - Diakonie Klinikum Dietrich Bonhoeffer, Neubrandenburg, Mecklenburg-Vorpommern
  - Klinikum Südstadt Rostock, Rostock, Mecklenburg-Vorpommern
  - Marien Kliniken, St. Marien-Krankenhaus, Siegen, Nordhein-Westfalen
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Städt. Kliniken Bielefeld gem. GmbH - Klinikum Mitte, Bielefeld, North Rhine-Westphalia
  - Augusta Kranken Anstalt Bochum, Bochum, North Rhine-Westphalia
  - Helios Klinikum Duisburg, Duisburg, North Rhine-Westphalia
  - Krankenhaus Düren gGmbH, Düren, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Klinikum Gütersloh, Gütersloh, North Rhine-Westphalia
  - St. Barbara-Klinik Hamm GmbH, Hamm, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Diakonie Klinikum GmbH Jung-Stilling-Krankenhaus, Siegen, North Rhine-Westphalia
  - Stiftungsklinikum Mittelrhein GmbH, Koblenz, Rhineland-Palatinate
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Klinikum St. Georg gGmbH, Leipzig, Saxony
  - Elblandkliniken Stiftung & Co.KG, Riesa, Saxony
  - Krankenhaus Martha-Maria Halle-Dölau, Halle, Saxony-Anhalt
  - Universitätsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Städtisches Krankenhaus Kiel GmbH, Kiel, Schleswig-Holstein
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Helios Klinikum Berlin-Buch, Berlin
  - Ev. Diakonie-Krankenhaus gemeinn. GmbH Bremen, Bremen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanoun M, Ruhnke L, Kramer M, Hanoun C, Schafer-Eckart K, Steffen B, Sauer T, Krause SW, Schliemann C, Mikesch JH, Kaufmann M, Hanel M, Jost E, Brummendorf TH, Fransecky L, Kraus S, Einsele H, Niemann D, Neubauer A, Kullmer J, Seggewiss-Bernhard R, Gorner M, Held G, Kaiser U, Scholl S, Hochhaus A, Reinhardt HC, Platzbecker U, Baldus CD, Muller-Tidow C, Bornhauser M, Serve H, Rollig C; Study Alliance Leukemia (SAL). Intensified cytarabine dose during consolidation in adult AML patients under 65 years is not associated with survival benefit: real-world data from the German SAL-AML registry. J Cancer Res Clin Oncol. 2023 Jul;149(8):4611-4621. doi: 10.1007/s00432-022-04356-9. Epub 2022 Sep 28. PMID 36167894
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Rollig C, Kramer M, Schliemann C, Mikesch JH, Steffen B, Kramer A, Noppeney R, Schafer-Eckart K, Krause SW, Hanel M, Herbst R, Kunzmann V, Einsele H, Jost E, Brummendorf TH, Scholl S, Hochhaus A, Neubauer A, Sohlbach K, Fransecky L, Kaufmann M, Niemann D, Schaich M, Frickhofen N, Kiani A, Heits F, Krumpelmann U, Kaiser U, Kullmer J, Wass M, Stolzel F, von Bonin M, Middeke JM, Thiede C, Schetelig J, Berdel WE, Ehninger G, Baldus CD, Muller-Tidow C, Platzbecker U, Serve H, Bornhauser M. Does time from diagnosis to treatment affect the prognosis of patients with newly diagnosed acute myeloid leukemia? Blood. 2020 Aug 13;136(7):823-830. doi: 10.1182/blood.2019004583. PMID 32496541
- See also: Website study alliance leukemia — https://www.aml-germany.com/register/aml-register